CLINICAL TRIAL: NCT04673539
Title: Adaptation and Validation of the Spanish Version of the Brief-BESTest in Stroke Patients
Brief Title: Spanish Version of the Brief-BESTest in Stroke Patients
Status: Completed | Type: Observational
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Inés Llamas-Ramos, Assistant Professor, University of Salamanca
Other Study IDs: NEUROUSAL01/2020
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Stroke
Keywords: Stroke; Validation Study; Postural Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group: Instrument validation in stroke patients
  Interventions: Diagnostic Test: Spanish version of the Brief-BESTest in stroke patients

INTERVENTIONS:
Diagnostic Test: Spanish version of the Brief-BESTest in stroke patients — Adaptation and validation of the Spanish version of the Brief-BESTest in stroke Patients

SUMMARY:
The aim of this study is to adapt and validate the Spanish version of the Brief-BESTest in stroke patients

DETAILED DESCRIPTION:
Balance disorder is a major risk factor for falls. The population that has suffered a cerebrovascular accident (CVA) or stroke has balance disorders. Over the last few years the assessment of balance has taken on special importance, carrying out the development, adaptation and validation of various tools that assess it.

The Brief-BESTest has 6 items, it has demonstrated comparable reliability to the Mini-BESTest and potentially superior sensitivity. This version represents all dimensions based on the original BESTest theory.

The purpose is to adapt and validate the Spanish version of the Brief-BESTest in stroke patients in order to have a brief tool, appropriate to the clinical environment and to the characteristics and limitations of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Diagnosis of stroke

Exclusion Criteria:

* Cognitive impairment
* Physical disability that prevents them from completing the assessment
* No cooperation and communication problems

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
BESTest | Baseline
Mini-BESTest | Baseline
Berg Balance Test | Baseline
Time Up and Go Test | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided